CLINICAL TRIAL: NCT05947474
Title: ORB-011 In Patients With Advanced Solid Tumors
Acronym: ORB
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Orionis Biosciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OR1-01
Record Dates: First submitted 2023-06-07; First posted 2023-07-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Cancer
Keywords: solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation ORB-011 (Experimental): ORB-011 Dose Escalation Participants will be administered study drug at dose levels corresponding to their Cohort. Cohort 1 will be treated with the lowest dose, and the dose will be escalated for future cohorts once the previous dose has been observed not to be associated with DLTs. Up to 7 dose cohorts have been pre-specified. Doses from the escalation arms will be selected as RP2D candidates.
  Interventions: Drug: ORB-011

INTERVENTIONS:
Drug: ORB-011 — Drug: ORB-011 is dosed via IV infusion

SUMMARY:
The goal of this clinical research study is to determine if an investigational new drug, named ORB-011, developed by Orionis Biosciences is safe and can be tolerated in people diagnosed with an advanced solid tumor.

The study also aims to find the biologically optimal dose of the study medicine by assessing the safety and potential activity in the treatment of solid tumors.

There are three phases to this study: screening, treatment and end of treatment.

DETAILED DESCRIPTION:
ORB-011 is a complex engineered biologic molecule that targets interferon alpha 2b activation specifically to type 1 conventional dendritic cells (cDC1). The interferon alpha 2b in ORB-011 is inactive to all other cell types but confers full activation in cis when bound to cDC1 cells which exclusively express CLEC9a, thereby eliminating the potential systemic toxicities caused by alpha interferon when binding to interferon receptors on other cells. ORB-1 is administered by intravenous (IV) infusion. In cancer patients, treatment may be repeated every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet the following criteria for inclusion:

  1. Age 18 years or older
  2. Patients with evidence of recurrent or refractory colorectal, HR+, triple-negative breast cancer (TNBC), non-small cell lung cancer (NSCLC), pancreatic cancer, head and neck squamous cell carcinoma (HNSCC), or metastatic melanoma, bladder/urothelial, gastric, esophageal, renal cell, hepatic, ovarian or other solid tumors deemed medically safe to undergo serial biopsies.
  3. Must have received or be ineligible for all standard of care therapies as deemed appropriate by the treating physician.
  4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
  5. Adequate organ and marrow function as defined below:

     * Hemoglobin ≥ 9.0 g/dL
     * Absolute neutrophil count (ANC) ≥ 1.5 × 109

       /L (> 1500 per mm3
     * Platelet count ≥ 75 × 109

       /L (> 75,000 per mm^3)
     * Serum bilirubin less than or equal to 1.5 × institutional upper limit of normal (ULN).
     * AST (SGOT)/ALT (SGPT) less than or equal to 2.5 × institutional ULN
     * Creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976)
     * Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 3 days prior to treatment. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (at least 12 consecutive months with no menses without an alternative medical cause)
  6. Patients and their partners must practice approved forms of contraception. Sexually active WCBP must agree to use a highly effective method of contraception prior to study entry and continuing for 30 days after ORB-011 administration. Highly effective methods of contraception are highly effective birth control methods with a failure rate of < 1% per year when used consistently and correctly. Additionally, male patients should refrain from donating sperm for 3 months following the last dose of study drug.
  7. Ability to understand and willingness to sign an Institutional Review Board (IRB)- approved written informed consent document (or that of legally authorized representative, if applicable)

Exclusion Criteria:

* Exclusion Criteria:

Patients are to be excluded from the study if they meet any of the following criteria:

1. Patients who are receiving any other investigational agents
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ORB-011 or its excipients.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

   Urinary tract infections (UTIs) are excluded from being an exclusion criterion for treatment unless they are Grade 3 or higher.
4. Pregnant women are excluded from this study because the effects of ORB-011 on a pregnant woman or fetus are unknown. Breastfeeding should be discontinued as the potential risk for AEs in nursing infants treated with ORB-011 is unknown.
5. Patients with hydronephrosis, except for those patients where hydronephrosis has been longstanding (ie, predates the diagnosis of the CIS, Ta, or T1 by more than 2 years) and diagnostic evaluation at screening shows no evidence of tumor causing the hydronephrosis
6. Any other anticancer therapy (eg, chemotherapy, biologic therapy, immunotherapy, targeted therapy, endocrine therapy, radiation therapy, intravesical therapy, investigational agent) within 28 days or 5 half-lives (whichever is shorter) of the study treatment
7. The patient has a diagnosis of another malignancy within 2 years before the first dose of study treatment, except for superficial skin cancer, localized prostate cancer on active surveillance, or localized solid tumors deemed cured by surgery and not treated with systemic anticancer therapy and not expected to require anticancer therapy in the next 2 years
8. Current or prior use of immunosuppressive medication within 28 days before ORB-011 treatment with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg. colitis or Crohn s disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism stable on hormonal replacement
   * Patients without active disease in the last 5 years may be included
   * Patients with celiac disease controlled by diet alone
10. History of primary immunodeficiency
11. History of allogeneic organ transplant
12. History of hypersensitivity to interferon alpha 2b or any excipient
13. Active infection with:

    * Tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and PPD testing if indicated),
    * Hepatitis B (HBV) or hepatitis C Virus (HBC): Patients with active HBV infection or active HCV infection are ineligible. However, patients with a history of HBV infection who have undetectable or low levels of HBV DNA and normal ALT are eligible. Patients with chronic HBV infection who meet the criteria for anti-HBV therapy are eligible if they have initiated anti-HBV therapy prior to treatment with ORB-011.

    Patients with a history of HCV infection are eligible if they have completed curative antiviral treatment and have a viral load that is below the limit of detection.
    * HIV: Patients living with HIV infection are ineligible only if they have a CD4 count less than 350 cells/µL and a history of an AIDS-defining infection within the last 12 months. Patients with a CD4 count greater than 350 cells/µL or who have not had an AIDS-defining infection within the last 12 months are eligible. Eligible patients living with HIV should maintain effective anti-retroviral therapy.
    * SARS-COV2 (PCR positive)
14. Receipt of live attenuated vaccination within 28 days prior to the study treatment
15. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
16. Patients with uncontrolled seizures
17. Any unresolved toxicity National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
18. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with ORB-011 may be included only after consultation with the Principal Investigator
19. Patients with QTcF > 480 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AE) in patients dosed with ORB-011 | 12 months
  Number of participants with adverse events (AE) in patients dosed with ORB-011
Determine Recommended Phase 2 Dose (RP2D) | 12 months
  Identify a RP2D for future studies.

SECONDARY OUTCOMES:
Measure Maximum Plasma Concentration [Cmax]). | 12 months
  Measure Maximum Plasma Concentration [Cmax]) of ORB-011 in patients
Collect the number of Dose Limiting Toxicities (DLTs) in patients dosed with ORB-001 | 12 months
  Record the number of DLTs

CONTACTS AND LOCATIONS:
Overall Officials: Robert Petit, PhD, Study Chair — SVP Early Clinical Development
Locations (2):
- United States (2):
  - Honor Health Research Institute, Scottsdale, Arizona
  - MD Anderson Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No